CLINICAL TRIAL: NCT07361328
Title: Low-intensity Ultrasonic Neuromodulation for Alleviation of Fibromyalgia Symptoms
Brief Title: Personalized Ultrasonic Brain Stimulation for Fibromyalgia
Acronym: BEAMforFMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Akiko Okifuji, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00188950
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia (FM)
Keywords: Fibromyalgia; Ultrasound brain stimulation; Clinical trials; MRI
MeSH Terms: conditions — Fibromyalgia | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Group (Experimental): Participants in this group will receive low-intensity ultrasound brain stimulation
  Interventions: Device: Low-intensity ultrasound brain stimulation
- Sham control (Sham Comparator): Participants in this group will undergo the same procedure with the Ultrasound group but do not receive ultrasound stimulation
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Low-intensity ultrasound brain stimulation — The device is called BEAM, which looks like an oversized pair of goggles that can be fitted over a participant's head. Once fastened, it emits a low-intensity ultrasound wave from your temples that targets a specific area of the brain. The treatment lasts about 45 minutes per session. In this study, participants will undergo a total of 6 sessions within a period of 2 weeks.
  Other Names: BEAM; Ultrasonic
  Arms: Ultrasound Group
Device: Sham (No Treatment) — There will be no ultrasound stimulation delivered
  Arms: Sham control

SUMMARY:
The primary purpose of this research is to evaluate a new kind of noninvasive brain stimulation intervention using the investigational ultrasound device, which might be useful for treating fibromyalgia. The device is for investigational use only and is not yet approved by the FDA for the intended use.

* Participants will be asked to visit the study center 7 times for in-person assessment and treatment sessions. In addition, participants will be asked to complete an online assessment 7 times. During in-person or online visits:

  * Participants will undergo an MRI scan twice during the first and last in-person visit (1 hour each) The second MRI may be optional.
  * There will be 6 treatment sessions (45 minutes each) within a 2-week period
* The online assessment occurs (15 minutes each)

  * two consecutive days before the first treatment session
  * 15 days after the first treatment session
  * 22 days after the first treatment session
  * 29 days after the first treatment session
  * 44 days after the first treatment session
  * 60 days after the first treatment session

DETAILED DESCRIPTION:
In this study, investigators will recruit 50 people with fibromyalgia. Participants will be asked to go through each of the following steps:

1. (In Person or Virtual) Initial visit (screening, medical history, questionnaires, 1 hour) 2. (Virtual) 2 daily pain ratings over two consecutive days (10 min each) 3. (In Person) MRI and 1st treatment session (MRI 1 hour, treatment 45 min, questionnaires 30 min) 4. (In Person) 4 treatment session visits (treatment 45 min each, questionnaires 30 min each) 5. (In Person) MRI (Optional) and last treatment session (MRI 1 hour, treatment 45 min, questionnaires 30 min) 6. (Virtual) questionnaires (20 min) 15 days after the first treatment session 7. (Virtual) questionnaires (20 min) 22 days after the first treatment session 8. (Virtual) questionnaires (20 min) 29 days after the first treatment session 9. (Virtual) questionnaires (20 min) 45 days after the first treatment session 10. (Virtual) questionnaires (20 min) 60 days after the first treatment session

1. Initial Visit In-person visit at the Pain Research Center or virtually, participants will be asked to complete a set of questionnaires designed to determine their health status, medical history, fibromyalgia-related symptoms, mood, and ability to do daily chores.

   Because pregnant women cannot participate in this study, study personnel will ask all female participants who have not achieved menopause to take a pregnancy test in person during this visit. If participants have a virtual visit, the pregnancy test will be done on the next in-person visit. Study personnel will escort participants to the bathroom, where participants will be given a small cup to collect urine. The urine sample will then be tested following the manufacturer's instructions to see if participants are pregnant.

   Once participants are deemed eligible, they will be assigned to either treatment or sham group. The assignment will be randomly determined at 1:1, meaning participants have 50/50 chance of being in treatment or sham group. If participants are in the Treatment group, they will receive low intensity ultrasound stimulation whereas if participants are in the Sham group, there will be no ultrasound emitted from the device.

   Study team will then schedule all treatment sessions. There will be a total of 6 treatment sessions within 2 weeks, and they must be separated by at least 24 hours.
2. Daily Pain Rating A few days before the MRI and first treatment session, study personnel will ask participants to rate their average and worst pain of the immediate past 24 hours once a day, for two consecutive days. Participants will receive a request on their phone or email to log into the University of Utah RedCap site to record the pain levels.
3. MRI and 1st Treatment Session Study personnel will meet participants at the University of Utah, Imaging & Neuroscience Center (729 Arapeen Drive) for the MRI session. Participants will be asked to remove all metal materials before being escorted into the MRI room. MRI creates images of the brain from magnetic signals. It does not use radiation. The MRI scan involves lying still on a table that moves into a hollow tunnel-like machine. The MRI technician will instruct participants to lie down on the table, stay awake and relaxed, and remain motionless during the scan.

   Before the MRI scan, participants will be asked to wear a flexible cap on their head to keep their hair down. The cap is a thin, flexible, MRI-compatible cap, similar to a swim cap. Study personnel will take two photos of their head from the side, one with the mock device (similar to the treatment device but without ultrasound) and the other without. Study personnel will provide participants with a surgical mask to wear for protection and privacy. After the pictures are taken, the research study staff will immediately perform the necessary calculations and blur the unmasked parts of their face. The original photographs will then be deleted. The photo-based calculation is needed for investigators to develop the ultrasound method that no longer requires MRI in the future.

   After the MRI, participants will receive the first ultrasound stimulation session. This will happen either in the private room at the Imaging & Neuroscience Center or participants will be asked to come to the Pain Research Center (a 6-minute walk or 2-minute drive). Participants will complete a questionnaire and receive the first treatment.

   Because this is a randomized clinical study, participants will be assigned to receive active, true ultrasound brain stimulation or sham stimulation. The procedure is the same for both. The study uses a device called BEAM. This is an investigational device that looks like an oversized pair of goggles that can be fitted over their forehead. Gel and mineral oil will be applied to each cup that will attach to the temples, and the device will be fastened. Participants will be seated comfortably during the session, which will last about 45 minutes. If participants are assigned to the treatment group, low intensity ultrasound will be emitted whereas if participants are assigned to the sham/placebo group, no ultrasound will be emitted. Once the device is removed, participants will be given a towel to clean the gel and oil. Participants will be asked to complete the questionnaire to rate their pain and mood.

   After each use, the cups that were attached to the temples will be removed and thoroughly cleaned with soap and warm water.
4. 2nd- 5th Treatment Session Participants will receive each treatment session at the Pain Research Center or Imaging & Neuroscience Center. The procedure is the same as the first treatment session. Additionally, participants will be asked to report any side effects from the treatment.
5. 6th Treatment Session and MRI Participants will receive the last (6th) treatment session at the Pain Research Center or Imaging & Neuroscience Center. The procedure is the same as the previous treatment session. Following this, participants may undergo the 2nd MRI scan at the Imaging & Neuroscience Center (optional). The procedure will be the same as the first MRI session.
6. Online Questionnaires Participants will be asked to complete the symptom questionnaires on

   * 15 days after the first treatment session
   * 22 days after the first treatment session
   * 29 days after the first treatment session
   * 45 days after the first treatment session
   * 60 days after the first treatment session Participants will receive a request notification on their phone or email to log into the University of Utah RedCap to complete the questionnaires. Each takes about 10-20 minutes.

The study participation will end after the last online questionnaire session.

ELIGIBILITY:
Inclusion Criteria:

* Meets American College of Rheumatology criteria for fibromyalgia:

  * Generalized pain, defined as pain in at least 4 of 5 regions, is present.
  * Widespread pain index (WPI) ≥ 7 and symptom severity scale score (SSS) ≥ 5, or WPI of 4-6 and SSS score ≥ 9.
  * Symptoms have been present at a similar level for at least 3 months.
  * d.A diagnosis of fibromyalgia is valid irrespective of other diagnoses. A diagnosis of fibromyalgia does not exclude the presence of other clinically important illnesses
* Failure of at least two evidence based medications (i.e., pregabalin, duloxetine, milnacipran) for the treatment of fibromyalgia.
* Failure of one or more attempts at physical therapy including:

  * Aerobic exercise like walking, cycling, and swimming,
  * Water therapy/hydrotherapy with warm water exercises,
  * Tai Chi involving slow, controlled movements,
  * Yoga,
  * Resistance training,
  * Bodyweight exercises,
  * Pilates,
  * Myofascial release therapy applying gentle pressure on trigger points,
  * Massage therapy,
  * Trigger point therapy targeting specific pain points,
  * Joint mobilization,
  * Postural retraining to correct body alignment,
  * Balance and coordination exercises,
  * Feldenkrais method for movement awareness,
  * Alexander technique to enhance posture and movement efficiency,
  * Transcutaneous Electrical Nerve Stimulation (TENS) for pain relief,
  * Heat therapy using hot packs, infrared, or paraffin wax,
  * Cold therapy with ice packs or cryotherapy,
  * Ultrasound therapy for deep tissue relaxation,
  * Biofeedback to control muscle tension and pain response,
  * Gentle static stretching for prolonged duration,
  * Active dynamic stretching for full range of motion,
  * Proprioceptive Neuromuscular Facilitation (PNF) stretching,
  * Hydrotherapy pool exercises,
  * Ai Chi (water-based Tai Chi),
  * Underwater treadmill therapy,
  * Graded motor imagery (GMI),
  * Mirror therapy to retrain brain-body connections,
  * Mindfulness-based stress reduction (MBSR) combining meditation and movement,
  * Cognitive-behavioral therapy
  * Gaze stabilization techniques for dizziness and disorientation
* Pain score of ≥ 4 on Numerical Rating Scale (NRS-11) at Screening visit.
* Pain score of ≥ 4 on Numerical Rating Scale (NRS-11) at Baseline visit.
* Stated willingness and ability to comply with all study procedures, to receive no additional interventions, and to remain on the same psychiatric treatment regimen (e.g., medication, psychotherapy) beginning at least one (1) month prior to screening and for the duration of the main study period unless a change in treatment is recommended or agreed upon by the site principal investigator.
* For participants of reproductive potential: negative urine or blood pregnancy test at screening; agreement to use a highly effective method of contraception (≤ 1% pregnancy rate) including tubal ligation, vasectomized partner, IUD or IUS (intrauterine device or system), or long-acting contraceptives (LARC).
* Willing and able to provide informed consent

Exclusion Criteria:

* Any previous diagnosis of bipolar disorder or schizophrenia-spectrum disorder during the participant's lifetime, according to Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-5) criteria.
* Diagnosis of moderate or severe alcohol or other substance use disorder in the past 6 months, according to DSM-5 criteria.
* Diagnosis of obsessive compulsive disorder and/or posttraumatic stress disorder in the past 30 days, according to DSM-5 criteria, and which is unstable in the clinical judgment of the investigator.
* Primary diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder in the past 3 months, according to DSM-5 criteria.
* Clinically significant neurodevelopmental, neurocognitive, or personality disorder, according to DSM-5 criteria.
* Moderate-High Risk of Suicide, according to the Columbia-Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent (i.e., answers YES to Question 3 and NO to Question 6 (Moderate Risk), or YES to Question 4, 5, or 6 (High Risk)), or in the clinical judgement of the site principal investigator (PI).

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale Pain +15days. 0 (no pain) - 10 (worst pain) | 15 days after the first treatment
  Pain score on the 0-10 scale at Day 15 following the first treatment

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised +15days. 0 (no impact) - 100 (severe impact) | 15 days after the first treatment
  Day15 Fibromyalgia Impact Questionnaire- Revised
Day15 PROMIS29 (Patient-Reported Outcomes Measurement Information System) Interference scale: (20 little/no interference) - 80 (very high interference) | 15 days after the first treatment
  PROMIS-29 (Patient-Reported Outcomes Measurement Information System - Pain interference subscale)
Response Rate 30% | 7 days after the first treatment
  At least 30% reduction in numerical pain score at Day 7
Patient Global Impression of Improvement (1 Very much better - 7 very much worse) | 15 days after the first treatment
  Patient's own assessment of how much symptoms are improved at Day 15
Numerical Rating Scale11 pain score Day 60 (0 No pain - 10 Worst pain) | 60 days after the first treatment
  Numerical pain score at Day 60
Day 15 Columbia suicide Severity Rating Scale (2 No/Low risk - 25 High risk) | 15 days after the first treatment
  Suicidality measured by the Columbia Suicide Severity Rating Scale at Day 15

OTHER OUTCOMES:
Day 15 Patient-Reported Outcomes Measurement Information System) other scales: (20 little/no problem ) - 80 (very high level of problem) | 15 days after the first treatment
  Scores of PROMIS 20 scales other than interference at Day 15
Day 15 Brief Pain Inventory - short form (BPI-S) 0 no pain - 10 pain as bad as you can imagine | 15 days after the first treatment
  Scores of BPI-S pain scales at Day 15
Day 60 Fibromyalgia Impact Questionnaire Revised. 0 (no impact) - 100 (severe impact) | 60 days after the first treatment
  Fibromyalgia Impact Questionnaire Revised scores at Day 60
Day 60 Brief Pain Inventory: 0 (no problem) - 10 (worst problem) | 60 days after the first treatment
  Brief Pain Inventory scores at Day 60
Day 60 Day15 PROMIS29 (Patient-Reported Outcomes Measurement Information System) All subscale: (20 little/no problem) - 80 (very high level of problem) | 60 days after the first treatment
  PROMIS scale scores (except Interference) at Day 60
Blinding and Group Assignment Assessment (How certain are you that you received active or sham treatment) 0 Completely certain for Sham treatment, 50 completely uncertain, 100 Completely certain for Active treatment | 15 days after the first treatment
  Patient belief on the group assignment (validity for blinding)

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah
Locations (1):
- Pain Research Center, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Riis TS, Lunt S, Kubanek J. MRI free targeting of deep brain structures based on facial landmarks. Brain Stimul. 2025 Jan-Feb;18(1):131-137. doi: 10.1016/j.brs.2024.12.1478. Epub 2025 Jan 3. PMID 39755367
- [Result] Riis TS, Feldman DA, Losser AJ, Okifuji A, Kubanek J. Noninvasive targeted modulation of pain circuits with focused ultrasonic waves. Pain. 2024 Dec 1;165(12):2829-2839. doi: 10.1097/j.pain.0000000000003322. Epub 2024 Jul 30. PMID 39073370